CLINICAL TRIAL: NCT02933164
Title: A Feasibility Trial to Evaluate the Senseonics Continuous Glucose Monitoring System in Canada
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0024
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

ARMS (1):
- Arms (Experimental): Evaluation of the effectiveness of modified Sensor designs on the longevity (up to 180 days) of the Senseonics Continuous Glucose Monitoring (CGM) System. The investigation will also evaluate safety of the Senseonics CGM System usage, while in the clinic and during home use.
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Effectiveness and safety of a Continuous Glucose Monitoring System

SUMMARY:
The purpose of this clinical investigation is to evaluate the effectiveness of modified Sensor designs on the longevity (up to 180 days) of the Senseonics Continuous Glucose Monitoring (CGM) System. The investigation will also evaluate safety of the Senseonics CGM System usage, while in the clinic and during home use.

ELIGIBILITY:
Inclusion Criteria:

Male and Female Subjects meeting all of the following inclusion criteria will be included in this study:

1. Subjects age ≥12 years
2. Clinically confirmed diagnosis of diabetes mellitus for ≥1 year
3. Subject has signed an informed consent form and is willing to comply with protocol requirements

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria at the time of screening will be excluded from this study:

1. Female subjects of childbearing capacity (defined as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study.
2. A condition preventing or complicating the placement, operation, or removal of the Sensor or wearing of transmitter, including upper extremity deformities or skin condition.
3. Symptomatic coronary artery disease; unstable angina; myocardial infarction, transient ischemic attack or stroke in the past 6 months; uncontrolled hypertension (systolic>160 mm Hg or diastolic >100 mm Hg at time of screening); current congestive heart failure; history of cardiac arrhythmia (benign PACs and PVCs allowed). Subjects with asymptomatic coronary artery disease (e,g, CABG, stent placement or angioplasty) may participate if negative stress test within 1 year prior to screening and written clearance from Cardiologist documented.
4. History of hepatitis B, hepatitis C, or HIV
5. Currently receiving (or likely to need during the study period):

   immunosuppressant therapy; chemotherapy; anticoagulant/antithrombotic therapy (excluding aspirin); glucocorticoids (excluding ophthalmic or nasal). This exclusion does include the use of inhaled glucocorticoids and the use of topical glucocorticoids (over sensor site only); antibiotic for chronic infection (e.g. osteomyelitis,endocarditis)
6. A condition requiring or likely to require magnetic resonance imaging (MRI)
7. Known topical or local anesthetic allergy
8. Known allergy to glucocorticoids
9. Any condition that in the investigator's opinion would make the subject unable to complete the study or would make it not in the subject's best interest to participate in the study. Conditions include but are not limited to psychiatric conditions, known current or recent alcohol abuse or drug abuse by subject history, a condition that may increase the risk of induced hypoglycemia or risk related to repeated blood testing. Investigator will supply rationale for exclusion
10. Participation in another clinical investigation (drug or device) within 2 weeks prior to screening or intent to participate during the study period
11. The presence of any other active implanted device (as defined further in protocol)
12. The presence of any other CGM sensor or transmitter located in upper arm (other location is acceptable)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
CGM Relative Difference to Laboratory Reference reported as MARD | 180 days
  Mean absolute relative difference (MARD) for paired Sensor and reference measurements through 180 days post-insertion for reference glucose values from 40-400 mg/dL will be calculated for comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- LMC Clinical Research Inc., Toronto, Ontario, Canada